CLINICAL TRIAL: NCT01708798
Title: A Prospective Randomized Placebo-controlled Study of the Effect of Eplerenone on Left Ventricular Diastolic Function in Women Receiving Anthracycline Therapy for Breast Cancer
Brief Title: Study of the Effect of Eplerenone on Heart Function in Women Receiving Anthracycline Chemotherapy for Breast Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H12-00185
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: Diastolic heart failure
MeSH Terms: conditions — Breast Neoplasms; Heart Failure, Diastolic | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): One tablet by mouth daily. If serum potassium level is <5.0 mmol/L at four weeks, increase to two tablets by mouth daily.
  If estimated glomerular filtration rate (eGFR) is between 30-49 ml per min per 1.73m2, initial dose is: one tablet by mouth every other day. If serum potassium level is <5.0 mmol/L at four weeks, increase to one tablet by mouth daily.
  Interventions: Drug: Placebo
- Eplerenone (Experimental): Eplerenone 25 mg tablet by mouth daily. If serum potassium level is <5.0 mmol/L at four weeks, increase to two 25 mg tablets by mouth daily.
  If estimated glomerular filtration rate (eGFR) is between 30-49 ml per min per 1.73m2, initial dose is: eplerenone 25 mg tablet by mouth every other day. If serum potassium level is <5.0 mmol/L at four weeks, increase to 25 mg tablet by mouth daily.
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone
  Other Names: Inspra
  Arms: Eplerenone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Doxorubicin and other anthracyclines are commonly used to treat breast cancer and other types of cancer. Unfortunately, they can cause heart muscle damage, resulting in scarring, abnormal contraction and relaxation, and heart failure symptoms. This side effect occurs more frequently at higher doses, and limits the total dose that can be given to cancer patients. Eplerenone is an oral medication that prevents or reverses heart damage in other disease states, and is commonly used to treat heart failure. This study will investigate the use of eplerenone to protect the heart from these harmful side effects of doxorubicin.

Few therapies have been shown to prevent heart damage in patients receiving anthracyclines. Small studies have suggested that other heart failure medications (ACE inhibitors, beta-blockers) may reduce the incidence of cardiac toxicity, but eplerenone and other drugs in its class (aldosterone antagonists) have not previously been studied. Eplerenone inhibits enzyme pathways that cause scarring of the heart, and animal studies suggest that anthracyclines cause damage through these same pathways.

This study aims to investigate whether eplerenone protects the heart from the harmful effects of doxorubicin chemotherapy. Specifically, it will measure the effect that eplerenone has on heart muscle relaxation. It will randomly assign women undergoing chemotherapy with doxorubicin to one of two groups: one group will receive eplerenone, and the other group will receive placebo (sugar) pills. The subjects will not know which type of pills they are taking. Heart muscle relaxation will be measured at baseline, after completion of chemotherapy (8-12 weeks), and after 6 months. There will also be various blood tests measured in the study subjects, to determine whether there might be certain blood tests that identify patients at particularly high risk of heart toxicity after doxorubicin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III breast cancer
* Scheduled to undergo treatment with doxorubicin-based chemotherapy regimen
* Able to provide informed consent

Exclusion Criteria:

* Use of anthracycline agents other than doxorubicin
* Baseline LVEF ≤50% by any modality (nuclear, echo, MRI)
* Atrial fibrillation or flutter
* Mitral valve disease (More than mild mitral stenosis or regurgitation, previous mitral valve replacement or repair)
* Inability to obtain adequate echo images for required analysis
* Hyperkalemia (K+ >5.0)
* Glomerular filtration rate (GFR) <30 ml/min/1.73m2
* Uncontrolled hypertension, defined as having a systolic blood pressure > 180 mmHg and/or a diastolic blood pressure >110 mmHg
* Symptomatic hypotension or systolic blood pressure <85 mmHg
* History of hypersensitivity to eplerenone or spironolactone
* Significant hepatic disease (e.g., previously documented positive serology for viral hepatitis) or aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >3 times the upper limits of normal
* Concomitant treatment with spironolactone, potassium-sparing diuretics, potassium supplements, or strong inhibitors of cytochrome P450 3A4 (CYP3A4) (i.e. ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir, nelfinavir)
* History of alcohol and/or any other drug abuse
* Women who are either pregnant, lactating or of childbearing potential and not using an acceptable method of contraception
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in average E' (averaged septal E' and lateral E') | 6 months
  The average early diastolic tissue velocity of the mitral valve annulus measured by tissue Doppler echocardiography (averaged velocities of the mitral annulus measured at the lateral edge and the septal edge)

SECONDARY OUTCOMES:
Development of worsening diastolic function | 6 months
  Development of worsening diastolic function, defined as a decline by at least one American Society of Echocardiography gradation of diastolic dysfunction
Development of worsening systolic function | 6 months
  Development of worsening systolic function, defined as a decline in LVEF of ≥10% to ≤50%
Change in septal E' | 6 months
  Change in early diastolic tissue velocity of the septal mitral annulus (E', measured by tissue Doppler echocardiography)
Change in lateral E' | 6 months
  Change in early diastolic tissue velocity of the lateral mitral annulus (E', measured by tissue Doppler echocardiography)
Change in E/E' | 6 months
  Change in the ratio of early diastolic mitral inflow velocity (E, measured by pulse wave Doppler echocardiography) to the average early diastolic tissue velocity of the mitral annulus (E', measured by tissue Doppler echocardiography)
Change in E/A | 6 months
  Change in the ratio of peak early diastolic mitral inflow velocity (E) to peak mitral inflow velocity during atrial systole (A), both measured by pulse wave Doppler echocardiography
Change in left atrial volume index | 6 months
  Change in the left atrial volume index, defined as the left atrial volume measured on the 2D echocardiogram indexed to body surface area
Change in left ventricular ejection fraction (LVEF) | 6 months
  Change in LVEF, measured by echocardiogram using Simpson's method
Biomarkers | Baseline, 1 week, 2 weeks, 4 weeks, 6 months
  Change in biomarkers of myocardial injury, inflammation, and collagen turnover as predictors of cardiotoxicity

OTHER OUTCOMES:
Incidence of hyperkalemia | 6 months
  Incidence of hyperkalemia defined as serum potassium >5.5 mmol/L
Incidence of adverse events leading to discontinuation of study drug | 6 months
  Incidence of adverse events leading to discontinuation of study drug, including hypotension, dizziness, hyperkalemia, or renal failure
Signal-averaged ECG (SAECG) changes | Baseline, 8-12 weeks, 6 months
  Change in late potentials measured on SAECG
Exercise stress test | Baseline, 6 months
  Change in QT/RR interval slope, exercise capacity, peak heart rate, heart rate recovery, ventricular arrhythmias during exercise, ventricular arrhythmias during recovery, presence of ischemia
Genetic predictors of cardiotoxicity and of response to eplerenone | 6 months
  Genetic predictors of cardiotoxicity and of response to eplerenone
ECG changes | Pre- and post-chemotherapy infusions (over 8-12 weeks)
  Change in QT interval, arrhythmias
Global longitudinal strain (GLS) | 6 months
  Change in GLS from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sean A Virani, MD, MSc, MPH, Principal Investigator — University of British Columbia; Margot Davis, MD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Cancer Agency, Vancouver Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Von Hoff DD, Layard MW, Basa P, Davis HL Jr, Von Hoff AL, Rozencweig M, Muggia FM. Risk factors for doxorubicin-induced congestive heart failure. Ann Intern Med. 1979 Nov;91(5):710-7. doi: 10.7326/0003-4819-91-5-710. PMID 496103
- [Background] Swain SM, Whaley FS, Gerber MC, Weisberg S, York M, Spicer D, Jones SE, Wadler S, Desai A, Vogel C, Speyer J, Mittelman A, Reddy S, Pendergrass K, Velez-Garcia E, Ewer MS, Bianchine JR, Gams RA. Cardioprotection with dexrazoxane for doxorubicin-containing therapy in advanced breast cancer. J Clin Oncol. 1997 Apr;15(4):1318-32. doi: 10.1200/JCO.1997.15.4.1318. PMID 9193323
- [Background] Wouters KA, Kremer LC, Miller TL, Herman EH, Lipshultz SE. Protecting against anthracycline-induced myocardial damage: a review of the most promising strategies. Br J Haematol. 2005 Dec;131(5):561-78. doi: 10.1111/j.1365-2141.2005.05759.x. PMID 16351632
- [Background] Kizaki K, Ito R, Okada M, Yoshioka K, Uchide T, Temma K, Mutoh K, Uechi M, Hara Y. Enhanced gene expression of myocardial matrix metalloproteinases 2 and 9 after acute treatment with doxorubicin in mice. Pharmacol Res. 2006 Apr;53(4):341-6. doi: 10.1016/j.phrs.2006.01.001. Epub 2006 Feb 7. PMID 16455267
- [Background] Goetzenich A, Hatam N, Zernecke A, Weber C, Czarnotta T, Autschbach R, Christiansen S. Alteration of matrix metalloproteinases in selective left ventricular adriamycin-induced cardiomyopathy in the pig. J Heart Lung Transplant. 2009 Oct;28(10):1087-93. doi: 10.1016/j.healun.2009.06.025. PMID 19782292
- [Background] Spallarossa P, Altieri P, Garibaldi S, Ghigliotti G, Barisione C, Manca V, Fabbi P, Ballestrero A, Brunelli C, Barsotti A. Matrix metalloproteinase-2 and -9 are induced differently by doxorubicin in H9c2 cells: The role of MAP kinases and NAD(P)H oxidase. Cardiovasc Res. 2006 Feb 15;69(3):736-45. doi: 10.1016/j.cardiores.2005.08.009. Epub 2005 Oct 6. PMID 16213474
- [Background] Zhao Y, McLaughlin D, Robinson E, Harvey AP, Hookham MB, Shah AM, McDermott BJ, Grieve DJ. Nox2 NADPH oxidase promotes pathologic cardiac remodeling associated with Doxorubicin chemotherapy. Cancer Res. 2010 Nov 15;70(22):9287-97. doi: 10.1158/0008-5472.CAN-10-2664. Epub 2010 Sep 30. PMID 20884632
- [Background] Clark JE, Sarafraz N, Marber MS. Potential of p38-MAPK inhibitors in the treatment of ischaemic heart disease. Pharmacol Ther. 2007 Nov;116(2):192-206. doi: 10.1016/j.pharmthera.2007.06.013. Epub 2007 Jul 24. PMID 17765316
- [Background] Bellahcene M, Jacquet S, Cao XB, Tanno M, Haworth RS, Layland J, Kabir AM, Gaestel M, Davis RJ, Flavell RA, Shah AM, Avkiran M, Marber MS. Activation of p38 mitogen-activated protein kinase contributes to the early cardiodepressant action of tumor necrosis factor. J Am Coll Cardiol. 2006 Aug 1;48(3):545-55. doi: 10.1016/j.jacc.2006.02.072. Epub 2006 Jul 12. PMID 16875982
- [Background] Martos R, Baugh J, Ledwidge M, O'Loughlin C, Conlon C, Patle A, Donnelly SC, McDonald K. Diastolic heart failure: evidence of increased myocardial collagen turnover linked to diastolic dysfunction. Circulation. 2007 Feb 20;115(7):888-95. doi: 10.1161/CIRCULATIONAHA.106.638569. Epub 2007 Feb 5. PMID 17283265
- [Background] Klappacher G, Franzen P, Haab D, Mehrabi M, Binder M, Plesch K, Pacher R, Grimm M, Pribill I, Eichler HG, et al. Measuring extracellular matrix turnover in the serum of patients with idiopathic or ischemic dilated cardiomyopathy and impact on diagnosis and prognosis. Am J Cardiol. 1995 May 1;75(14):913-8. doi: 10.1016/s0002-9149(99)80686-9. PMID 7733000
- [Background] Host NB, Jensen LT, Bendixen PM, Jensen SE, Koldkjaer OG, Simonsen EE. The aminoterminal propeptide of type III procollagen provides new information on prognosis after acute myocardial infarction. Am J Cardiol. 1995 Nov 1;76(12):869-73. doi: 10.1016/s0002-9149(99)80251-3. PMID 7484822
- [Background] Di Zhang A, Nguyen Dinh Cat A, Soukaseum C, Escoubet B, Cherfa A, Messaoudi S, Delcayre C, Samuel JL, Jaisser F. Cross-talk between mineralocorticoid and angiotensin II signaling for cardiac remodeling. Hypertension. 2008 Dec;52(6):1060-7. doi: 10.1161/HYPERTENSIONAHA.108.117531. Epub 2008 Nov 3. PMID 18981328
- [Background] Hori Y, Yoshioka K, Kanai K, Hoshi F, Itoh N, Higuchi S. Spironolactone decreases isoproterenol-induced ventricular fibrosis and matrix metalloproteinase-2 in rats. Biol Pharm Bull. 2011;34(1):61-5. doi: 10.1248/bpb.34.61. PMID 21212518
- [Background] Rude MK, Duhaney TA, Kuster GM, Judge S, Heo J, Colucci WS, Siwik DA, Sam F. Aldosterone stimulates matrix metalloproteinases and reactive oxygen species in adult rat ventricular cardiomyocytes. Hypertension. 2005 Sep;46(3):555-61. doi: 10.1161/01.HYP.0000176236.55322.18. Epub 2005 Jul 25. PMID 16043662
- [Background] Zannad F, Dousset B, Alla F. Treatment of congestive heart failure: interfering the aldosterone-cardiac extracellular matrix relationship. Hypertension. 2001 Nov;38(5):1227-32. doi: 10.1161/hy1101.099484. PMID 11711528
- [Background] Zannad F, Alla F, Dousset B, Perez A, Pitt B. Limitation of excessive extracellular matrix turnover may contribute to survival benefit of spironolactone therapy in patients with congestive heart failure: insights from the randomized aldactone evaluation study (RALES). Rales Investigators. Circulation. 2000 Nov 28;102(22):2700-6. doi: 10.1161/01.cir.102.22.2700. PMID 11094035
- [Background] Jensen BV, Skovsgaard T, Nielsen SL. Functional monitoring of anthracycline cardiotoxicity: a prospective, blinded, long-term observational study of outcome in 120 patients. Ann Oncol. 2002 May;13(5):699-709. doi: 10.1093/annonc/mdf132. PMID 12075737
- [Background] Marchandise B, Schroeder E, Bosly A, Doyen C, Weynants P, Kremer R, Pouleur H. Early detection of doxorubicin cardiotoxicity: interest of Doppler echocardiographic analysis of left ventricular filling dynamics. Am Heart J. 1989 Jul;118(1):92-8. doi: 10.1016/0002-8703(89)90077-x. PMID 2741800
- [Background] Ewer MS, Ali MK, Mackay B, Wallace S, Valdivieso M, Legha SS, Benjamin RS, Haynie TP. A comparison of cardiac biopsy grades and ejection fraction estimations in patients receiving Adriamycin. J Clin Oncol. 1984 Feb;2(2):112-7. doi: 10.1200/JCO.1984.2.2.112. PMID 6699662
- [Background] Dodos F, Halbsguth T, Erdmann E, Hoppe UC. Usefulness of myocardial performance index and biochemical markers for early detection of anthracycline-induced cardiotoxicity in adults. Clin Res Cardiol. 2008 May;97(5):318-26. doi: 10.1007/s00392-007-0633-6. Epub 2008 Jan 14. PMID 18193371
- [Background] Di Lisi D, Bonura F, Macaione F, Peritore A, Meschisi M, Cuttitta F, Novo G, D'Alessandro N, Novo S. Chemotherapy-induced cardiotoxicity: role of the tissue Doppler in the early diagnosis of left ventricular dysfunction. Anticancer Drugs. 2011 Jun;22(5):468-72. doi: 10.1097/CAD.0b013e3283443704. PMID 21301318
- [Background] Nagy AC, Cserep Z, Tolnay E, Nagykalnai T, Forster T. Early diagnosis of chemotherapy-induced cardiomyopathy: a prospective tissue Doppler imaging study. Pathol Oncol Res. 2008 Mar;14(1):69-77. doi: 10.1007/s12253-008-9013-4. Epub 2008 Mar 15. PMID 18347931
- [Background] Pudil R, Horacek JM, Strasova A, Jebavy L, Vojacek J. Monitoring of the very early changes of left ventricular diastolic function in patients with acute leukemia treated with anthracyclines. Exp Oncol. 2008 Jun;30(2):160-2. PMID 18566583
- [Background] Tassan-Mangina S, Codorean D, Metivier M, Costa B, Himberlin C, Jouannaud C, Blaise AM, Elaerts J, Nazeyrollas P. Tissue Doppler imaging and conventional echocardiography after anthracycline treatment in adults: early and late alterations of left ventricular function during a prospective study. Eur J Echocardiogr. 2006 Mar;7(2):141-6. doi: 10.1016/j.euje.2005.04.009. Epub 2005 Jun 6. PMID 15941672
- [Background] Nagueh SF, Sun H, Kopelen HA, Middleton KJ, Khoury DS. Hemodynamic determinants of the mitral annulus diastolic velocities by tissue Doppler. J Am Coll Cardiol. 2001 Jan;37(1):278-85. doi: 10.1016/s0735-1097(00)01056-1. PMID 11153752
- [Background] Hayashi SY, Rohani M, Lindholm B, Brodin LA, Lind B, Barany P, Alvestrand A, Seeberger A. Left ventricular function in patients with chronic kidney disease evaluated by colour tissue Doppler velocity imaging. Nephrol Dial Transplant. 2006 Jan;21(1):125-32. doi: 10.1093/ndt/gfi075. Epub 2005 Oct 12. PMID 16221719
- [Background] Kasner M, Westermann D, Steendijk P, Gaub R, Wilkenshoff U, Weitmann K, Hoffmann W, Poller W, Schultheiss HP, Pauschinger M, Tschope C. Utility of Doppler echocardiography and tissue Doppler imaging in the estimation of diastolic function in heart failure with normal ejection fraction: a comparative Doppler-conductance catheterization study. Circulation. 2007 Aug 7;116(6):637-47. doi: 10.1161/CIRCULATIONAHA.106.661983. Epub 2007 Jul 23. PMID 17646587
- [Background] Edwards NC, Ferro CJ, Kirkwood H, Chue CD, Young AA, Stewart PM, Steeds RP, Townend JN. Effect of spironolactone on left ventricular systolic and diastolic function in patients with early stage chronic kidney disease. Am J Cardiol. 2010 Nov 15;106(10):1505-11. doi: 10.1016/j.amjcard.2010.07.018. PMID 21059444
- [Background] Vizzardi E, D'Aloia A, Giubbini R, Bordonali T, Bugatti S, Pezzali N, Romeo A, Dei Cas A, Metra M, Dei Cas L. Effect of spironolactone on left ventricular ejection fraction and volumes in patients with class I or II heart failure. Am J Cardiol. 2010 Nov 1;106(9):1292-6. doi: 10.1016/j.amjcard.2010.06.052. Epub 2010 Sep 9. PMID 21029826
- [Background] Mottram PM, Haluska B, Leano R, Cowley D, Stowasser M, Marwick TH. Effect of aldosterone antagonism on myocardial dysfunction in hypertensive patients with diastolic heart failure. Circulation. 2004 Aug 3;110(5):558-65. doi: 10.1161/01.CIR.0000138680.89536.A9. Epub 2004 Jul 26. PMID 15277317
- [Background] Pitt B, Remme W, Zannad F, Neaton J, Martinez F, Roniker B, Bittman R, Hurley S, Kleiman J, Gatlin M; Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study Investigators. Eplerenone, a selective aldosterone blocker, in patients with left ventricular dysfunction after myocardial infarction. N Engl J Med. 2003 Apr 3;348(14):1309-21. doi: 10.1056/NEJMoa030207. Epub 2003 Mar 31. PMID 12668699
- [Background] Zannad F, McMurray JJ, Krum H, van Veldhuisen DJ, Swedberg K, Shi H, Vincent J, Pocock SJ, Pitt B; EMPHASIS-HF Study Group. Eplerenone in patients with systolic heart failure and mild symptoms. N Engl J Med. 2011 Jan 6;364(1):11-21. doi: 10.1056/NEJMoa1009492. Epub 2010 Nov 14. PMID 21073363
- [Background] Pinto JT, Delman BN, Dutta P, Nisselbaum J. Adriamycin-induced increase in serum aldosterone levels: effects in riboflavin-sufficient and riboflavin-deficient rats. Endocrinology. 1990 Sep;127(3):1495-501. doi: 10.1210/endo-127-3-1495. PMID 2387263
- [Background] Cardinale D, Sandri MT. Role of biomarkers in chemotherapy-induced cardiotoxicity. Prog Cardiovasc Dis. 2010 Sep-Oct;53(2):121-9. doi: 10.1016/j.pcad.2010.04.002. PMID 20728699
- [Background] Jensen BV, Nielsen SL, Skovsgaard T. Treatment with angiotensin-converting-enzyme inhibitor for epirubicin-induced dilated cardiomyopathy. Lancet. 1996 Feb 3;347(8997):297-9. doi: 10.1016/s0140-6736(96)90469-9. PMID 8569365
- [Background] Georgakopoulos P, Roussou P, Matsakas E, Karavidas A, Anagnostopoulos N, Marinakis T, Galanopoulos A, Georgiakodis F, Zimeras S, Kyriakidis M, Ahimastos A. Cardioprotective effect of metoprolol and enalapril in doxorubicin-treated lymphoma patients: a prospective, parallel-group, randomized, controlled study with 36-month follow-up. Am J Hematol. 2010 Nov;85(11):894-6. doi: 10.1002/ajh.21840. PMID 20872550
- [Background] Seidman A, Hudis C, Pierri MK, Shak S, Paton V, Ashby M, Murphy M, Stewart SJ, Keefe D. Cardiac dysfunction in the trastuzumab clinical trials experience. J Clin Oncol. 2002 Mar 1;20(5):1215-21. doi: 10.1200/JCO.2002.20.5.1215. PMID 11870163